CLINICAL TRIAL: NCT06039865
Title: Augmenting Obstructive Sleep Apnea Chronic Care Management With Consumer Wearable Devices in Patients Prescribed Positive Airway Pressure Therapy
Brief Title: Chronic Care Management With Wearable Devices in Patients Prescribed Positive Airway Pressure Therapy (mPAP) Trial
Acronym: mPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Constance Fung, Principal Investigator, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20233750
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Wearable; Pulse oximetry; Sleep apnea; Treatment adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Participants will be provided with a consumer wearable immediately after randomization to wear for 4 weeks.
  Interventions: Behavioral: Immediate Intervention
- Waitlist control (Other): Participants will receive usual care from the sleep center for 6 weeks and then be provided with a consumer wearable to wear for 4 weeks.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Immediate Intervention — Participants will receive customized weekly reports from the pulse oximetry data collected by the consumer wearable.
  Arms: Immediate Intervention
Behavioral: Waitlist control — Participants only receive usual care from the sleep center.
  Arms: Waitlist control

SUMMARY:
The goal of this clinical trial in adults with obstructive sleep apnea prescribed positive airway pressure therapy is to test the effects of a new patient-facing consumer wearable-based program (that involves provision of a consumer wearable that measures oxygen levels during sleep plus customized weekly reports to participants). The main question is to learn whether participants' use of positive airway pressure therapy will differ between the participants who receive the new program immediately versus delayed. Participants assigned to the delayed program will receive usual care while waiting for the program to begin.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomized to immediate versus waitlist control in a 1:1 ratio.

Our project is at the forefront of consumer wearable research, leveraging the recent capabilities of consumer wearables to provide pulse oximetry data during sleep, to uncover new ways to promote PAP usage among patients with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed PAP therapy from the sleep center for > 1 week
* Have an active profile in our Center's ResMed AirView or Respironics Care Orchestrator accounts for > 1 week
* Non-adherent with PAP therapy
* Willing to continue using current PAP device for 28 days continuously
* Have an electronic device compatible with the wearable app

Exclusion Criteria:

* Diagnosis of heart failure, chronic lung disease, dementia, active substance use disorder
* Use home oxygen
* Unstable medical or psychiatric illness
* Planned non-use of PAP therapy (e.g., waiting for replacement of recalled PAP device)
* Planned surgery or hospitalization during study period
* Planned extensive travel during study period
* History of repeated non-attendance at clinic visits

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
PAP adherence (minutes) | 5 weeks
  Change in mean minutes of PAP use per night between baseline (T1) and post-treatment (T3).

SECONDARY OUTCOMES:
PAP adherence (percent of days used >= 4 hours) | 5 weeks
  Change in the percent of days PAP was used >= 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Constance H. Fung, MD, MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA Greater Los Angeles Healthcare System, North Hills, California, United States

REFERENCES:
- [Derived] Mak S, Ash G, Liang LJ, Der-McLeod E, Ghadimi S, Kewalramani A, Naeem S, Zeidler M, Fung C. Testing a Consumer Wearables Program to Promote the Use of Positive Airway Pressure Therapy in Patients With Obstructive Sleep Apnea: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 19;13:e60769. doi: 10.2196/60769. PMID 39207912